CLINICAL TRIAL: NCT06662188
Title: A Phase 1/2, Multicenter, Open-Label, Dose-Escalation, Safety, Tolerability, and Clinical Activity Study of a Single Dose of JAG201 Gene Therapy Delivered Via Intracerebroventricular Administration in Participants With SHANK3 Haploinsufficiency
Brief Title: JAG201 Gene Therapy Study in Children & Adults With SHANK3 Haploinsufficiency
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jaguar Gene Therapy, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAG-201-CL-101
Record Dates: First submitted 2024-10-16; First posted 2024-10-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: SHANK3 Haploinsufficiency; Phelan-McDermid Syndrome
Keywords: SHANK3 Haploinsufficiency; SHANK3; Phelan-McDermid Syndrome
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, first-in-human (FIH), single-dose, dose-escalation, safety, tolerability, and clinical activity of JAG201. A traditional 3+3 design strategy will be implemented for dose escalation from the 1st cohort to the 2nd cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pediatric Cohort 1 (Experimental): Starting Dose
- Pediatric Cohort 2 (Experimental): Escalated Dose
  Interventions: Genetic: JAG201

INTERVENTIONS:
Genetic: JAG201 — Adeno-associated virus 2/9 expressing a miniature version of the human SHANK3 gene (AAV2/9-miniSHANK3)
Genetic: JAG201 — Adeno-associated virus 2/9 expressing a miniature version of the human SHANK3 gene (AAV2/9-miniSHANK3)
  Arms: Pediatric Cohort 2

SUMMARY:
This is a Phase 1/2, first in human, open-label, dose-escalation study to evaluate the safety, tolerability, and clinical activity of a single dose of JAG201 administered via intracerebroventricular (ICV) injection in pediatric and adult participants with SHANK3 haploinsufficiency resulting from SHANK3 loss of function mutations and chromosomal deletions encompassing the SHANK3 gene. Clinical data will be evaluated for safety, tolerability, and preliminary clinical activity of JAG201 in pediatric and adult participants with SHANK3 haploinsufficiency. The pediatric cohorts will start enrolling first and the enrollment for adult cohorts may be initiated at a later timepoint in the study.

DETAILED DESCRIPTION:
A target of 6 pediatric participants aged 2 to 9 years will be treated in Cohorts 1 and 2. In total, all participants will be followed for safety and tolerability for at least 5 years after the date of treatment with JAG201. The study will include 5 periods: Pre-Screening, Screening, Gene Therapy Administration and Perioperative Management, Initial Follow-Up, and Long-Term Follow-Up. Study participants will be evaluated for treatment eligibility during the Pre-Screening and Screening Periods. The Pre-Screening/Screening Period may be up to 90 days before treatment with JAG201 (Day 1). On Day 1, treatment-eligible participants will receive a one-time ICV injection of JAG201. Participant safety will be monitored closely after JAG201 administration in a hospital setting. During the Initial Follow-Up Period, up to Year 2, participants will return at regularly scheduled intervals for safety and clinical activity assessments. Participants will continue the study in the Long-Term Follow-Up Period through Year 5.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is male or female, and 2 to 9 years of age at the time of JAG201 administration
2. Has a molecular confirmation of a loss of function mutation in SHANK3 or a 22q13.3 deletion classified as a Class I deletion
3. Has evidence of developmental/cognitive delay of at least 2 standard deviations (SD) below the mean (i.e., ≤ 70) via either Intelligence Quotient (IQ) OR Developmental Quotient (DQ) assessment (as applicable)
4. Has an overall Phelan-McDermid Syndrome (PMS) Assessment of Severity (PMSA-S) Score of 3 or greater at Screening
5. Willing to initiate structured therapies and continue for the duration of the study as determined by the specific therapist (structured therapies may include, at a minimum, physical therapy, occupational therapy, speech therapy, and applied behavior analysis)
6. Is stable on any medication regimens (if being administered to control the signs and symptoms of underlying disease) for at least 3 months prior to the planned JAG201 study treatment
7. If undergoing any kind of behavioral or therapeutic intervention, then the level of intervention must have remained stable for at least 3 months prior to the planned JAG201 study treatment (exclusive of school vacations/illness).
8. Is a permanent legal resident of the U.S. residing within the continental U.S.

Key Exclusion Criteria:

A pediatric participant who meets any of the following criteria will be excluded from this study:

1. Has history of developmental regression defined in this study as a prolonged loss of previously acquired skills (defined as skills maintained for at least 3 months) with loss of skills persisting for at least 3 months
2. Has known or suspected prion disease (e.g., Creutzfeldt-Jakob Disease)
3. Has poorly-controlled epilepsy (defined as an increase in the dose or addition of new anti-epileptic medications within the past 3 months) or any history of status epilepticus or seizure-induced hospitalizations within the last 12 months
4. Has history of acute cerebrovascular episodes
5. Has active autoimmune disease or prior treatment with immunomodulatory therapy, immunotherapy, and/or immunosuppressive drugs within 3 months prior to study enrollment (Note: Inhaled or topical steroids are permitted in the absence of active autoimmune disease)
6. Has infection (viral, bacterial, or fungal) that requires treatment < 6 weeks before JAG201 administration (Note: JAG201 administration may be postponed until the infection has resolved and the participant is clinically stable)
7. Has medical illness or other concern that would cause the Investigator to conclude that the participant will not be able to perform the study procedures or assessments or would confound interpretation of data obtained during assessments
8. Has known allergy or hypersensitivity to prednisolone or other glucocorticosteroids, or their excipients
9. Has received any vaccine < 6 weeks before JAG201 administration
10. Has received any gene therapy

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-01-07 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Enrollment to Month 60
  Incidence, type, severity, and frequency of AEs
Incidence of Serious Adverse Events (SAEs) | Enrollment to Month 60
  Incidence, type, severity, and frequency of SAEs
Clinically significant abnormalities in laboratory values | Enrollment to Month 60
  Changes in clinically significant abnormalities in laboratory values
Incidence of immunogenicity response abnormalities | Enrollment to Month 60
  Incidence of anti-AAV9 antibodies, anti-transgene antibodies, and T-cell reactivity to transgene over time

SECONDARY OUTCOMES:
Change from Baseline in SAND | Enrollment to Month 60
  To characterize the preliminary disease response to JAG201 by assessing the change from baseline in SAND (Sensory Assessment for Neurodevelopmental Disorders)

OTHER OUTCOMES:
Change from baseline in Vineland Adaptive Behavior Scales | Enrollment to Month 60
  To characterize further the preliminary clinical activity of JAG201 by assessing change from baseline in Vineland Adaptive Behavior Scales, Third Edition

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gallo, PhD, Study Director — Jaguar Gene Therapy
Locations (3):
- United States (3):
  - Rush University, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Seaver Autism Center at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No